CLINICAL TRIAL: NCT06906081
Title: Finerenone Treatment for Diabetic Cardiovascular Autonomic Neuropathy: the FibroCAN Study
Acronym: FibroCAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peter Rossing (Other)
Collaborators: Steno Diabetes Center Nordjylland (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Peter Rossing, MD, professor, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-516597-30-00; 2024-516597-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-03; First posted 2025-04-02 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Autonomic Neuropathy; Type 2 Diabetes; Diabetic Neuropathies
Keywords: Mineralocorticoid receptor antagonist (MRA); Cardiovascular autonomic neuropathy; Type 2 Diabetes; Diabetic Neuropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies | interventions — finerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Finerenone (active) (Experimental)
  Interventions: Drug: Kerendia (Finerenone, BAY94-8862)

INTERVENTIONS:
Drug: Kerendia (Finerenone, BAY94-8862) — Titration of finerenone will be based on baseline eGFR. Participants with eGFR > 60 mL/min/1.73m² will start on a 20mg dosage. Medication dosage will be increased to 40 mg after one month if serum potassium < 4.8 mmol/l. If side effects occur at any dosage, the dosage will be reduced to the previous level.
  Participants with eGFR < 60 and >25 Participants with eGFR < 60 mL/min/1.73m² (and eGFR < 25 mL/min/1.73m²) will start on a 10mg dosage. Medication dosage will be increased to 20 mg after one month if serum potassium < 4.8 mmol/l. Subsequently, Medication dosage will be increased to 40 mg after an additional one month if serum potassium < 4.8 mmol/l. If side effects occur at any dosage, the dosage will be reduced to the previous level.
  Finerenone is administered orally as immediate release tablets.
  Arms: Finerenone (active)
Drug: Placebo — Placebo tablets matching BAY94-8862 are administered orally.
  Arms: Placebo

SUMMARY:
Diabetic neuropathy is a serious and common complication of diabetes that currently has no cure. One form of this condition is cardiovascular autonomic neuropathy (CAN), which affects about 20% of people with diabetes-an estimated 100 million people worldwide. CAN is a significant risk factor for death and health problems like heart disease and kidney damage, and may contribute to the high rates of cardiovascular-related deaths in people with diabetes.

This study is a double-blind, randomized, placebo-controlled, two-center trial. The study aims to test whether finerenone can treat cardiovascular autonomic neuropathy in patients with type 2 diabetes. The trial will evaluate the effects of 78 weeks of treatment with finerenone or a placebo, assigned randomly in a 1:1 ratio, on early-stage cardiovascular autonomic neuropathy. The trial will include 100 participants with type 2 diabetes. Additionally, the study will investigate how the treatment impacts other types of neuropathy and related pathological mechanisms.

ELIGIBILITY:
To be included in this study the participants must fulfill the following inclusion criteria.

* Given informed consent
* Type 2 diabetes defined by WHO criteria
* Aged 40 ≥ at inclusion
* Pathological E/I ratio (Mean value of three measures)

Exclusion criteria Participants will be excluded in one or more of the following criteria are met.

* No CAN (no abnormal CARTs)
* Definite CAN (more than one abnormal CART)
* HbA1C >100 mmol/L
* Treatment with potassium-sparing diuretics (amiloride) or MRAs e.g., spironolactone or eplerenone which cannot be discontinued 4 weeks prior to screening visit. The patient's primary physician, who is not involved in this study, will determine if discontinuation is possible.
* Atrial fibrillation/flutter
* Congestive heart failure (NYHA class 3-4)
* History of cardiac arrhythmia
* Severe forms of respiratory disease including asthma and COPD
* Any nondiabetic cause of neuropathy
* All female subjects of childbearing potential (WOCBP) must have a negative result of a highly sensitive urine HCG (pregnancy test) performed at screening. Subjects of childbearing potential must agree to use a highly effective form of contraception throughout the duration of the study (list of definition on WOCBP and accepted contraception in appendix A).
* Severe hepatic impairment
* Lactose intolerance
* Breastfeeding
* Nephropathy requiring dialysis
* Beta-blocker-use
* Hyperkalemia at screening visit (plasma potassium >4.8 mmol/l)
* eGFR < 25 ml/min/1.73m2
* Potassium plasma > 4.8 mmol/l (at randomization)
* Treatment with strong CYP3A4-inhibitors (e.g. Itraconazol, ketoconazol, ritonavir, cobicistat, clarithromycin) which cannot be discontinued 4 weeks prior to screening visit
* Treament with moderate to strong CYP3A4-induceres (e.g. rifampicin, carbamazepine, phenytoin, phenobarbital, St John's Wort or efavirenz) which cannot be discontinued 4 weeks prior to screening visit
* Have received chemotherapeutic treatment within last 12 months
* Grapefruit consumption that cannot be discontinued during the study period
* Inability to complete study protocol, assessed to investigator
* Not able to read, write and/or understand Danish

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Between-group (finerenone vs. placebo) difference in changes on the CART E/I ratio | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Measured by vagus device

SECONDARY OUTCOMES:
Between-group (finerenone vs. placebo) difference in changes on the CART R/S ratio | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  R/S ratio (CART). Measured by Vagus device.
Between-group (finerenone vs. placebo) difference in changes on the CART Valsalva manoeuvre. | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Valsalva manoeuvre (CART). Measured by Vagus device.
Between-group (finerenone vs. placebo) differences in changes on heart rate variability (HRV) by SDNN and RMSSD | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Measured by vagus device as SDNN (Standard Deviation of Normal-to-Normal interbeat) intervals and RMSSD (Root Mean Square of Successive Differences between normal heartbeats). SDNN and RMSSD is measured in milliseconds.
Between-group (finerenone vs. placebo) differences in changes on heart rate variability (HRV) by high and low frequency power. | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Measured by vagus device as low and high frequency power in the unit milliseconds squared.
Between-group (finerenone vs. placebo) differences in changes on fibrosis markers in serum | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78. Skin biopsies on week 0, week 36 and week 78.
  Serum PRO-C6 and PRO-C3 assessed by ELISA.
Between-group (finerenone vs. placebo) differences in changes on fibrosis markers in skin biopsies by PRO-C6 | From baseline to the end of treatment at 78 weeks. Tested at week 0, 36 and 78
  Pro-C6 by immunostaining
Between-group (finerenone vs. placebo) differences in changes on fibrosis markers in skin biopsies by C3M | From baseline to the end of treatment at 78 weeks. Tested at week 0, 36 and 78
  C3M by immunostaining

OTHER OUTCOMES:
Between-group (finerenone vs. placebo) differences in changes on inflammation markers | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Olink inflammation markers will be measured with PCR.
Between-group (finerenone vs. placebo) differences in changes on markers of retinopathy | From enrollement to the end of treatment at 78 weeks. Tested at week 0, week 36 and week 78.
  Markers of retinopathy (nonproliferativ/proliferative retinopathy and retinal nerve fibre layer thickness by optical coherence tomography)
Between-group (finerenone vs. placebo) differences in changes on markers of corneal neuropathy by CNFD | From enrollement to the end of treatment at 78 weeks. Tested at week 0, week 36 and week 78.
  Overall to quantify the severity of small nerve fibre damage by confocal corneal microscopy. Quantified by corneal nerve fiber density (CNFD) measured in fibers per mm2.
Between-group (finerenone vs. placebo) differences in changes on markers of corneal by neuropathy by CNBD | From enrollement to the end of treatment at 78 weeks. Tested at week 0, week 36 and week 78.
  Overall to quantify the severity of small nerve fibre damage by confocal corneal microscopy.
  Quantified including corneal nerve branch density (CNBD) measured in branches per mm2.
Between-group (finerenone vs. placebo) differences in changes on markers of corneal neuropathy by DCF, DCP, NCF and NCP | From enrollement to the end of treatment at 78 weeks. Tested at week 0, week 36 and week 78.
  Overall to quantify the severity of small nerve fibre damage by confocal corneal microscopy. Quantified including corneal nerve fiber length (CNFL), dendritic cells with contact to nerve fiber (DCF), dendritic cells without contact to nerve fiber (DCP), non-dendritic cells with contact to nerve fiber (NCF) and non-dendritic cells without contact to nerve fiber (NCP). All measured in cells per mm2.
Between-group (finerenone vs. placebo) difference on Cardiac vagal tone | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Measured with eMotion Faros
Between-group (finerenone vs. placebo) difference in changes on questionnaires for painful and painless neuropathy DN4 | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  The following neuropathy questionnaires will be used to assess peripheral neuropathy:
  - The Douleur Neuropathique 4 (DN4) to assess painful peripheral neuropathy with a cut-off ≥ 4.
Between-group (finerenone vs. placebo) difference in changes on questionnaires for painful and painless neuropathy MNSI | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  The following neuropathy questionnaires will be used to assess peripheral neuropathy:
  Michigan Neuropathy Screening Instrument (MNSI) with ≥ 4 a cut-off.
Between-group (finerenone vs. placebo) difference in changes on orthostatic blood pressure testing | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Orthostatic hypotension will be defined as decline in systolic blood pressure ≥ 20 mmHg or diastolic blood pressure ≥ 10 mmHg or a decrease in systolic blood pressure to < 90. From position change from lying to standing.
Between-group (finerenone vs. placebo) difference in changes on Sudomotor function of the skin in hands and feet (Sudoscan) | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Measured with: (Sudoscan)
Between-group (finerenone vs. placebo) difference in changes of questionnaires for autonomic neuropathy Compass-31 | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Measured with compass-31.
Between-group (finerenone vs. placebo) difference in changes of questionnaires for autonomic neuropathy GCSI | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Measured with GCSI.
Between-group (finerenone vs. placebo) difference in changes of sural nerve conduction and amplitude (DPNCheck) | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Nerve conduction velocity and amplitude of the sural nerve will be assessed the average of three measures on both the left and right leg by use of the NC-StatR DPNCheck (NeuroMetrix, Inc., Waltham, USA). Age- and height-stratified perception thresholds will be applied.
Between-group (finerenone vs. placebo) difference in changes of vibration sensation threshold (Biothesiometry) | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Vibration perception threshold (VPT) will be measured by using biothesiometry (Bio-medical instruments, Ohio, USA) applied to the distal tip of the first toe on both feet. Cut-off above 25 V and age-sex-height specific cut-offs was applied (38, 39). Biothesiometry measurements will be repeated three times and averaged of the measures will be used.
Between-group (finerenone vs. placebo) difference in changes of pain sensation | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Pain sensation will be assessed by pinprick (Neuropen, Owen Mumford Ltd, Oxford, UK). Pinpricks will be applied proximal to the nail on the first dorsal, third and fifth toes on each foot. DPN will be defined as no pain at any tested location.
Between-group (finerenone vs. placebo) difference in changes of light touch sensation | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Ten-gram monofilament (Neuropen, Owen Mumford Ltd, Oxford, UK) will be applied three times at four points on the plantar aspect of the foot (first toe, proximal to the first toe, third toe and fifth toe) in addition to the proximal to the nail on the first dorsal, third and fifth toes on each foot. All measures will be obtained on both feet. DPN will be defined as absence of sensation at all locations.
Between-group (finerenone vs. placebo) difference in changes of cold and warm sensation of foot and lower leg | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Thermal sensation (25°C and 40°C) will be assessed by applying metal rolls bilaterally on the dorsal side of the first toe, dorsum of the foot and the anterior part of the low leg from 10 centimeter above the lateral malleolus and 10 centimeter proximately by Rolltemp-II (Somedic SenseLab AB). All measures will be obtained on both legs. Abnormal sensation will be defined as bilateral abnormalities at the toes, either with or without an abnormal sensation of the foot and leg.
Between-group (finerenone vs. placebo) difference in changes of ancle and patella reflexes (Reflex hammer) | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 12, week 24, week 36, week 52 and week 78
  Ancle and patella reflexes will be perform using a reflex hammer on both sides.
Between-group (finerenone vs. placebo) difference in changes of intraepidermal nerve fiber density (IENFD) | From baseline to the end of treatment at 78 weeks. Tested at screening, week 0, week 36 and week 78
  Intraepidermal nerve fiber density (IENFD quantified following international guidelines
The association between serum fibrosis markers and level of peripheral neuropathy in type 2 diabetes | Data analysis after baseline sampling
  Measurement of baseline fibrosis markers in serum and in skin samples and compare to level of peripheal neuropathy measured at baseline
The association between serum fibrosis markers and level of autonomic neuropathy in type 2 diabetes | Data analysis after baseline sampling
  Measurement of baseline fibrosis markers in serum and compare to level of autonomic neuropathy measured at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, Professor, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (2):
- Denmark (2):
  - Steno Diabetes Center Northern Denmark, Gistrup
  - Steno Diabetes Center Copenhagen, Herlev

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Bitsch Poulsen M, Okdahl T, Buciek JH, Drewes AM, Karlsson P, Ahluwalia TS, Brock B, Brock C, Rossing P, Hansen CS. Protocol for the FibroCAN study: a randomised controlled trial of finerenone treatment for early-stage cardiovascular autonomic neuropathy in type 2 diabetes. BMJ Open. 2025 Oct 23;15(10):e101074. doi: 10.1136/bmjopen-2025-101074. PMID 41130701

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/81/NCT06906081/Prot_SAP_000.pdf